CLINICAL TRIAL: NCT06314919
Title: A Multicenter, Prospective, Cohort Study to Evaluate the Efficacy and Safety of Fixed-Dose Combination of Pitavastatin/Ezetimibe Under the Real-World Condition
Brief Title: A Study to Evaluate the Efficacy and Safety of Fixed-Dose Combination of Pitavastatin/Ezetimib
Status: Recruiting | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-PEC-OS-401
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Primary Hypercholesterolemia; Mixed Dyslipidemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of fixed-Dose combination of Pitavastatin/Ezetimibe under the real-world condition

ELIGIBILITY:
Inclusion Criteria:

* Those who taking statins or statins and ezetimibe in addition to dietary and exercise therapy for primary hypercholesterolemia or mixed hyperlipidemia
* Those who are judged to need administration of a fixed-dose combination of pitavastatin/ezetimibe for change of statin's formulation or change of statin's dose, addition of ezetimibe

Exclusion Criteria:

* Those who are taking a fixed-dose combination of pitavastatin/ezetimibe at study enrollment
* Those with hypersensitivity reactions or relevant medical history to pitavastatin or ezetimibe
* Those who have been administered an investigational product within 12 weeks of the enrollment date or are planning to participate in another clinical trial during this study participation period.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who require administration of a fixed-dose combination of pitavastatin/ezetimibe for the treatment of primary hypercholesterolemia or mixed dyslipidemia
Sampling Method: Non-Probability Sample
Enrollment: 8606 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of reaching the target LDL Cholesterol level | 12 weeks after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Ewha Womans University Seoul Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No